CLINICAL TRIAL: NCT06325800
Title: The Role of Glycoxidation on Arterial Biomechanics and Target Organ Damage in Patients With Moderate to High Cardiovascular Risk. The GlycOxiTod Observational Multicentric Registry
Brief Title: Glycoxidation, Arterial Biomechanics, and Target Organ Damage
Acronym: GlycOxiTod
Status: Recruiting | Type: Observational
Sponsor: Complejo Hospitalario Universitario de Santiago (Other)
Collaborators: Instituto de Investigación Sanitaria de Santiago de Compostela (Unknown); Instituto de Salud Carlos III (Other Government); University of Santiago de Compostela (Other); Hospital de Barbanza (Unknown)
Responsible Party: Principal Investigator, Nestor Vazquez Agra, Principal Investigator, Complejo Hospitalario Universitario de Santiago
Other Study IDs: 2021401/2023007; Grant (Other Grant/Funding Number: Juan Rodés Grant (JR23/00018))
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Oxidative Stress; Cardiovascular Risk; Target Organ Damage
Keywords: glycation; antioxidant; target organ damage; arterial biomechanic; carotid; glycoxidation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — blood (plasma, serum), urine, salive, skin (no invasive)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Patients with
  Arterial biomechanics values lower than or equal to the 50th percentile of the distribution (measured as carotid stiffness by ultrasound elastography, distensibility and stress, flow velocity and vascular resistance),
  AND
  Absence of vascular target organ damage (considered as carotid intima-media thickness >0.9 mm, cholesterol plaque, carotid stenosis, carotid-femoral pulse wave velocity >10 m/s, pulse pressure >60 mmHg, ankle-Brachial Index <0.9 or >1.3, hypertensive retinopathy)
  AND
  Absence of cardiovascular disease (cardiovascular events, cerebrovascular events, hospital admissions, consultations, death, disability)
- Cases: Patients with
  Arterial biomechanics values higher than the 50th percentile of the distribution (measured as carotid stiffness by ultrasound elastography, distensibility and stress, flow velocity and vascular resistance),
  OR
  Presence of vascular target organ damage (considered as carotid intima-media thickness >0.9 mm, cholesterol plaque, carotid stenosis, carotid-femoral pulse wave velocity >10 m/s, pulse pressure >60 mmHg, ankle-Brachial Index <0.9 or >1.3, hypertensive retinopathy)
  OR
  Presence of cardiovascular disease (cardiovascular events, cerebrovascular events, hospital admissions, consultations, death, disability)

SUMMARY:
Vascular target organ damage (TOD), defined as structural or functional deleterious changes in large and small arteries, is related to unfavorable arterial biomechanics, atherosclerosis and arteriosclerosis. Endothelial dysfunction due to unfavorable redox and glycation states on the bases of these phenomena. However, little is known about the role of glycoxidation on arterial biomechanics and TOD in apparently healthy individuals. The main hypothesis is that glycation and glycoxidation status are associated with arterial biomechanical abnormalities and TOD in patients with moderate to high cardiovascular risk. This is an observational, ambispective, and multicenter project that will include non-smoking patients over 18 years, without diabetes mellitus or established cardiovascular disease. Demographic, epidemiological, and clinical-anthropometric variables will be collected, including data from ambulatory blood pressure monitoring. The investigators will measure the serum percentage of glycated hemoglobin, glycated albumin, and fructosamine levels; along with quantification of skin advanced glycation and glycoxidation end productos (AGEs). Plasma concentration, activity, and structure of catalase, glutathione peroxidase, and superoxide dismutase in relation to the patient's glycation and glycoxidation status will be also evaluated. Concurrently, several biomechanical parameters will be assessed in the Common, Internal Carotid Artery, and distal limb arteries using ultrasound exploration. Incipient microvasculature damage will be also evaluated by retinal image. Patients will be followed up for the development of arterial biomechanical abnormalities and TOD, along with cardiovascular events.

DETAILED DESCRIPTION:
INTRODUCTION

Atherosclerotic cardiovascular disease (ASCVD) represents one of the leading causes of morbidity and mortality in the population. Arterial hypertension (AHT), along with other cardiovascular risk (CVR) factors, predisposes to abnormalities in the structure and function of large and small arteries, leading to premature vascular aging and culminating in the development of target organ damage (TOD),which reresents a clear but underdiagnosed precursor of ASCVD. However, not all patients develop TOD, nor do they do so over the same time span or with the same intensity. Additionally, patients who initially present with low to moderate CVR are already considered to be at moderate to high CVR in the presence of TOD, with more stringent therapeutic objectives.

Vascular biomechanics primarily focuses on the study of mechanical properties and behavior of arteries. Unfavorable arterial biomechanics are associated with the development and progression of atherosclerosis and arteriosclerosis. These processes represent a continuum of vascular damage mediated by the accumulation of oxidized lipoproteins in the subendothelial space, activation and amplification of inflammatory pathways, and development of arterial fibrosis and calcification. At the core of these phenomena lies the occurrence of endothelial dysfunction, characterized by increased permeability and loss of the vascular endothelium's filtering capacity for deleterious molecules to the arterial wall.

Oxidative stress, defined as an imbalance between reactive species production and antioxidant systems in favor of the former, plays a crucial role in the development of endothelial dysfunction, deposition of oxidized lipoproteins, and proinflammatory interaction between these and the mononuclear-phagocytic system. The accumulation of reactive oxygen species (ROS) and others induces lipid peroxidation and glycoxidation phenomena culminating in the formation of advanced lipoxidation and glycation end products (ALEs and AGEs, respectively). ALEs and AGEs can bind to proteins, causing functional and structural abnormalities, and also influence cellular signaling by activating, among others, death pathways.

Unfavorable redox status and glycation levels are linked to aging, degenerative diseases, and accumulated vascular damage in certain subpopulations, particularly patients with diabetes mellitus (DM). However, little is known about the influence of antioxidant system glycation and glycoxidation on arterial biomechanics and the development of target organ damage in apparently healthy patients with moderate to high CVR. The investigators aim to study the specific relationship between arterial biomechanical abnormalities and TOD with serum glycation levels, glycoxidation status, and function-structure balance of some antioxidant system elements, highlighting catalase, superoxide dismutase, and glutathione peroxidase.

MATERIALS AND METHODS

Project Design and Setup

This is an observational, ambispective, and multicenter project promoted by the Unit of Hypertension and Cardiovascular risk belonging to the Internal Medicine Department at the University Hospital of Santiago de Compostela. Participants will be individuals belonging to the Organizational Structure of Integrated Management (EOXI) of Santiago de Compostela and Barbanza who seek consultation for CVR diagnosis, management, and follow-up.

Participants. Inclusion and Exclusion Criteria

From the total pool of consulted patients, only individuals over 18 years with a moderate to high CVR profile based on guideline reference scores will be preselected. Exclusion criteria will include the presence of DM according to current clinical practice guidelines, smoking habit (defined as current consumption and within the 6 months prior to recruitment), risky alcohol consumption (defined as consumption exceeding 10 g and 20 g daily for women and men, respectively), and established cardiovascular disease.

Assessment of Arterial Biomechanical Markers and TOD

The investigators will perform bilateral ultrasound exploration of the Common Carotid Artery (CCA), Internal Carotid Artery (ICA) and distal arteries of the lower limbs using a Mindray Z60 device (Mindray®, Guangdong, China) with high-frequency probe. The following measurements and calculations will be extracted:

1. In motion mode (M-mode), concomitant measurement of arterial radius, arterial pressures, and total wall thickness for the calculation of distensibility and tension parameters in the middle segment of the CCA.
2. In two-dimensional mode (B-mode), automated measurement of intima-media thickness (IMT) in the distal region of the CCA, along with detection and characterization of cholesterol plaque.
3. In spectral Doppler mode, morphological description of volume-time (flow) function in terms of flow velocities and vascular resistance indices in the middle segment of the CCA and ICA.
4. In B-mode with elastography module, direct evaluation of local stiffness degree in a middle segment of the CCA.
5. In spectral Doppler mode with ECG synchronization, assessment of carotid-femoral pulse wave velocity (c-f PWV).
6. In spectral Doppler mode, assessment of the ankle-brachial index (ABI).

The investigators will also assess incipient damage in the retinal microvasculature using retinography with a Topcon TRC-NW6S device (Electronics®, Tokyo, Japan).

Assessment of Oxidative Stress markers and Antioxidant System Activity-Structure

To assess the redox status, plasma and urine thiobarbituric acid reactive substances (TBARS) and reduced thiols will be assessed according to the referenced protocols via spectrophotometric quantification. Enzymatic function of glutathione peroxidase, catalase, and superoxide dismutase will be measured as enzymatic activity according to the referenced protocols. These analyses will be conducted using an Asys UVM-340 analyzer (Biochrom®, Cambridge, UK). Structure features of antioxidant enzymes based on glycation and glycoxidation patterns will be assessed using proteomics.

Determination of Glycation, Glycoxidation, and Lipoxidation status

The percentage of glycated hemoglobin will be assessed using high-performance liquid chromatography (HPLC) with the Hemoglobin next analyzer (A. Menarini Diagnostics®, Florence, Italy). Fructosamine levels will be determined by the diazyme glycated serum protein enzymatic method (Diazyme, Kent, UK) on an Advia 2400 analyser (Siemens Healthcare Diagnostics Inc.®, Tarrytown, USA). The percentage of glycated albumin will be estimated from fructosamine and albumin levels. This laboratory assessment will be performed by the Central Hospital Laboratory department.

General levels of glycoxidation and lipoxidation will be estimated through quantification of dicarbonyl levels using the TBARS spectrophotometric approach. Global glycoxidation status will be also estimated through assessment of skin advanced glycation end products (AGEs) using an AGE Reader (DiagnOptics BV®, Groningen, Netherlands). AGEs mainly represent glycated adducts bound to proteins that arise during glycoxidation processes. The AGE Reader has been developed to assess skin autofluorescence (SAF) non-invasively using the fluorescent properties of various AGEs.

Outcomes in Cardiovascular Risk

The investigators will measure the number needed to treat (NNT) of consultations and exploration time to detect abnormalities in arterial biomechanics and target organ damage (TOD), and thus determine an increased CVR warranting therapeutic intensification. Cardiovascular and cerebrovascular events, hospital admissions, consultations, death and disability will be also assessed.

Ethical Considerations and Good Clinical Practice

This study will be conducted in accordance with the ethical principles of the Declaration of Helsinki and the good practice standards in the research of the Galician (Spain) Health Service (SERGAS). Written informed consent will be obtained from all patients who agreed to participate. The protocols were approved by the Research Ethics Committee of Santiago-Lugo (codes 2021/401 and 2023/302).

Work Plan and Project Flow

In a first phase, the investigators plan to include patients meeting the criteria and consenting to participate. Clinical-anthropometric evaluation, arterial biomechanics, TOD detection, and sample collection will be conducted in a single medical act. Biomechanical, oxidative stress, glycation and glycoxidation markers will be quantified in both patients with and without biomechanical abnormalities and arterial TOD. The aim of this phase is to evaluate the differences between patient groups based on biomechanical parameters and arterial TOD. In a subgroup of patients, differences in the structure-function of antioxidant enzymes in terms of glycation and glycoxidation levels, and their relationship with arterial biomechanical abnormalities and TOD will also be evaluated. This phase will include the extraction, collection, processing, and analysis of preliminary data, along with the attainment of the project's initial results.

In a second phase,

1. Patients without biomechanical abnormalities or TOD will undergo a 5-year follow-up, with anual and final evaluations of biomechanical abnormalities, TOD, and cardiovascular outcomes. The aim of this phase is to evaluate differences in the previous markers between patient groups based on biomechanical parameters and arterial TOD. In a subgroup of patients, differences in the structure-function of antioxidant enzymes in terms of glycation and glycoxidation levels, and their relationship with arterial biomechanical abnormalities and TOD will be also assessed. This phase will include the extraction, collection, processing, and analysis of preliminary data, along with the attainment of the project's final results.
2. Patients with biomechanical abnormalities and/or TOD will undergo a 5-year follow-up, with annual and final evaluations of TOD progression and cardiovascular outcomes. The aim of this phase is to evaluate differences in the previous markers between patient groups based arterial TOD and cardiovascular outcomes. In a subgroup of patients, differences in the structure-function of antioxidant enzymes in terms of glycation and glycoxidation levels, and their relationship with TOD and cardiovascular outcomes will be assessed. This phase will include the extraction, collection, processing, and analysis of preliminary data, along with the attainment of the project's final results.

Mathematical analysis and modeling

The SPSS 22.0 statistical software package (SPSS Inc.®, Chicago, IL, EE.UU) will be employed. A descriptive statistic approach will be performed, including assessment of normality for quantitative variables. Univariate statistics will be used to compare groups with specific tests depending on the variable type. If relevant results are found, linear correlation studies will be conducted. After univariate analysis, multivariate models will be constructed, both explanatory for the association of predictors with the outcomes, and predictive for the risk of biomechanical abnormalities, TOD and cardiovascular results. To assess factors that may influence biomechanical parameters, TOD and cardiovascular results over time, specific mathematical procedures related to joint modeling approach and time series analysis will be applied. Sample size calculations will be based on specific statistical tests according to the variable type and distribution, always considering a moderate effect size, 95% confidence interval (95%CI), and at least 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Moderate to high Cardiovascular Risk estimated by SCORE2OP.
* Signed written consent for participation in the study.

Exclusion Criteria:

* Absence of current smoking habit and in the last 6 months.
* High-risk alcohol consumption (More than 10 and 20 g/day in women and men, respectively).
* Presence of Diabetes mellitus.
* Established cardiovascular disease, including heart failure, ischemic heart disease, valvular heart disease, atrial fibrillation, peripheral artery disease, and cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients belonging to the health area of Santiago de Compostela and Barbanza (A Coruña, Spain), referred from primary care and hospital services to the Cardiovascular Risk and Hypertension Unit of the Internal Medicine Department at the reference hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of redox status (1) | Present, two, four years and final (5 years)
  Evaluation of thiobarbituric acid reactive substances (TBARS) levels as a measure of lipid peroxidation
Assessment of redox status (2) | Present, two, four years and final (5 years)
  Evaluation of reduced thiol levels as a measure of protein oxidation
Evaluation of glycation status (1) | Present, two, four years and final (5 years)
  Measurement of serum fructosamine and glucose levels
Evaluation of glycation status (2) | Present, two, four years and final (5 years)
  Measurement of the percentage of serum glycated hemoglobin
Evaluation of glycation status (3) | Present, two, four years and final (5 years)
  Estimation of the percentage of serum glycated albumin
Evaluation of glycation status (4) | Present, two, four years and final (5 years)
  Quantification of skin advanced glycation end products (AGEs)
Assessment of Glycoxidation status (1) | Present, two, four years and final (5 years)
  Levels of thiobarbituric acid reactive substances (TBARS) also as an estimation of dicarbonyl levels from glycoxidation
Assessment of Glycoxidation status (2) | Present, two, four years and final (5 years)
  Quantification of skin advanced glycation end products (AGEs) also as an estimation of the levels of some glycoxidation byproducts
Quantification of arterial targen organ damage (TOD) during the follow-up (1) | Present, two, four years and final (5 years)
  Number of patients and severity (Arterial TOD considered as carotid intima-media thickness >0.9 mm, cholesterol plaque, carotid stenosis, carotid-femoral pulse wave velocity >10 m/s, pulse pressure >60 mmHg, ankle-Brachial Index <0.9 or >1.3 hypertensive retinopathy)
Quantification of arterial targen organ damage (TOD) during the follow-up (2) | two, four years and final (5 years)
  Number needed to treat (NNT) of consultations and exploration time to detect abnormalities in arterial biomechanics and target organ damage (TOD)

SECONDARY OUTCOMES:
Evaluation of cardiovascular disease during the follow-up | two, four years and final (5 years)
  Number of patients developing cardiovascular and cerebrovascular events, number of hospital admissions and consultations, number of patients with a cardiovascular fatal event, number of patients with disabilities and their degree of disability

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Background] Wang MC, Lloyd-Jones DM. Cardiovascular Risk Assessment in Hypertensive Patients. Am J Hypertens. 2021 Jun 22;34(6):569-577. doi: 10.1093/ajh/hpab021. PMID 33503227
- [Background] Piskorz D. Hypertensive Mediated Organ Damage and Hypertension Management. How to Assess Beneficial Effects of Antihypertensive Treatments? High Blood Press Cardiovasc Prev. 2020 Feb;27(1):9-17. doi: 10.1007/s40292-020-00361-6. Epub 2020 Jan 23. PMID 31975151
- [Background] Simon BR, Kaufmann MV, McAfee MA, Baldwin AL. Finite element models for arterial wall mechanics. J Biomech Eng. 1993 Nov;115(4B):489-96. doi: 10.1115/1.2895529. PMID 8302030
- [Background] Guzik TJ, Touyz RM. Oxidative Stress, Inflammation, and Vascular Aging in Hypertension. Hypertension. 2017 Oct;70(4):660-667. doi: 10.1161/HYPERTENSIONAHA.117.07802. Epub 2017 Aug 7. No abstract available. PMID 28784646
- [Background] Vistoli G, De Maddis D, Cipak A, Zarkovic N, Carini M, Aldini G. Advanced glycoxidation and lipoxidation end products (AGEs and ALEs): an overview of their mechanisms of formation. Free Radic Res. 2013 Aug;47 Suppl 1:3-27. doi: 10.3109/10715762.2013.815348. PMID 23767955
- [Background] Gianazza E, Brioschi M, Fernandez AM, Banfi C. Lipoxidation in cardiovascular diseases. Redox Biol. 2019 May;23:101119. doi: 10.1016/j.redox.2019.101119. Epub 2019 Feb 25. PMID 30833142
- [Background] Al-Kuraishy HM, Sami OM, Hussain NR, Al-Gareeb AI. Metformin and/or vildagliptin mitigate type II diabetes mellitus induced-oxidative stress: The intriguing effect. J Adv Pharm Technol Res. 2020 Jul-Sep;11(3):142-147. doi: 10.4103/japtr.JAPTR_18_20. Epub 2020 Jul 14. PMID 33102198
- [Background] Mattson MP. Roles of the lipid peroxidation product 4-hydroxynonenal in obesity, the metabolic syndrome, and associated vascular and neurodegenerative disorders. Exp Gerontol. 2009 Oct;44(10):625-33. doi: 10.1016/j.exger.2009.07.003. Epub 2009 Jul 19. PMID 19622391
- [Background] Hospital Clínico Universitario de Santiago - Área Sanitaria de Santiago de Compostela y Barbanza (Hospitales, Centros de Salud, Casas del Mar y Consultorios) n.d. https://xxisantiago.sergas.es/Paxinas/web.aspx? tipo=paxtab&idLista=3&idContido=183&migtab=174%3B183&idioma=es (accessed March 12, 2024).
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Briasoulis A, Agarwal V, Messerli FH. Alcohol consumption and the risk of hypertension in men and women: a systematic review and meta-analysis. J Clin Hypertens (Greenwich). 2012 Nov;14(11):792-8. doi: 10.1111/jch.12008. Epub 2012 Sep 25. PMID 23126352
- [Background] Amos A, Greaves L, Nichter M, Bloch M. Women and tobacco: a call for including gender in tobacco control research, policy and practice. Tob Control. 2012 Mar;21(2):236-43. doi: 10.1136/tobaccocontrol-2011-050280. Epub 2011 Dec 13. PMID 22166266
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S19-S40. doi: 10.2337/dc23-S002. PMID 36507649
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Diaz-Louzao C, Barrera-Lopez L, Lopez-Rodriguez M, Casar C, Vazquez-Agra N, Pernas-Pardavila H, Marques-Afonso A, Vidal-Vazquez M, Montoya JG, Andrade AH, Fernandez-Castro I, Varela P, Gonzalez-Quintela A, Otero E, Gude F, Cadarso-Suarez C, Tome S. Longitudinal relationship of liver injury with inflammation biomarkers in COVID-19 hospitalized patients using a joint modeling approach. Sci Rep. 2022 Apr 1;12(1):5547. doi: 10.1038/s41598-022-09290-x. PMID 35365705
- [Background] Malone HE, Nicholl H, Coyne I. Fundamentals of estimating sample size. Nurse Res. 2016 May;23(5):21-5. doi: 10.7748/nr.23.5.21.s5. PMID 27188569
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. New York: Routledge; 1988. https://doi.org/10.4324/9780203771587.
- [Result] Bozkurt Yilmaz HE, Yilmaz M. Assessment of Carotid Artery Distensibility and Elasticity in Patients with Asthma. Iran J Allergy Asthma Immunol. 2021 Jun 6;20(3):279-286. doi: 10.18502/ijaai.v20i3.6329. PMID 34134449
- [Result] Strandberg TE, Pitkala K. What is the most important component of blood pressure: systolic, diastolic or pulse pressure? Curr Opin Nephrol Hypertens. 2003 May;12(3):293-7. doi: 10.1097/00041552-200305000-00011. PMID 12698068
- [Result] Molinari F, Zeng G, Suri JS. A state of the art review on intima-media thickness (IMT) measurement and wall segmentation techniques for carotid ultrasound. Comput Methods Programs Biomed. 2010 Dec;100(3):201-21. doi: 10.1016/j.cmpb.2010.04.007. Epub 2010 May 15. PMID 20478640
- [Result] Andrikou I, Tsioufis C, Konstantinidis D, Kasiakogias A, Dimitriadis K, Leontsinis I, Andrikou E, Sanidas E, Kallikazaros I, Tousoulis D. Renal resistive index in hypertensive patients. J Clin Hypertens (Greenwich). 2018 Dec;20(12):1739-1744. doi: 10.1111/jch.13410. Epub 2018 Oct 25. PMID 30362245
- [Result] Sigrist RMS, Liau J, Kaffas AE, Chammas MC, Willmann JK. Ultrasound Elastography: Review of Techniques and Clinical Applications. Theranostics. 2017 Mar 7;7(5):1303-1329. doi: 10.7150/thno.18650. eCollection 2017. PMID 28435467
- [Result] Ji H, Xiong J, Yu S, Chi C, Bai B, Teliewubai J, Lu Y, Zhang Y, Xu Y. Measuring the Carotid to Femoral Pulse Wave Velocity (Cf-PWV) to Evaluate Arterial Stiffness. J Vis Exp. 2018 May 3;(135):57083. doi: 10.3791/57083. PMID 29781986
- [Result] Zwakenberg SR, de Jong PA, Hendriks EJ, Westerink J, Spiering W, de Borst GJ, Cramer MJ, Bartstra JW, Doesburg T, Rutters F, van der Heijden AA, Schalkwijk C, Schurgers LJ, van der Schouw YT, Beulens JWJ; SMART Study Group. Intimal and medial calcification in relation to cardiovascular risk factors. PLoS One. 2020 Jul 13;15(7):e0235228. doi: 10.1371/journal.pone.0235228. eCollection 2020. PMID 32658909
- [Result] Ohkawa H, Ohishi N, Yagi K. Assay for lipid peroxides in animal tissues by thiobarbituric acid reaction. Anal Biochem. 1979 Jun;95(2):351-8. doi: 10.1016/0003-2697(79)90738-3. No abstract available. PMID 36810
- [Result] ELLMAN GL. Tissue sulfhydryl groups. Arch Biochem Biophys. 1959 May;82(1):70-7. doi: 10.1016/0003-9861(59)90090-6. No abstract available. PMID 13650640
- [Result] Aebi H. Catalase in vitro. Methods Enzymol. 1984;105:121-6. doi: 10.1016/s0076-6879(84)05016-3. No abstract available. PMID 6727660
- [Result] Flohe L, Gunzler WA. Assays of glutathione peroxidase. Methods Enzymol. 1984;105:114-21. doi: 10.1016/s0076-6879(84)05015-1. No abstract available. PMID 6727659
- [Result] Kwas M, Bucholc B, Slusarczyk J. [Use of electrophoresis in polyacrylomide gel (SDS_PAGE) for evaluating IgG structure--the main component of human intravenous immunoglobulin]. Med Dosw Mikrobiol. 2000;52(3):301-9. Polish. PMID 11147272
- [Result] Chaila MZ, Viniegra M, Gagliardino JJ, Martinez A, Simesen de Bielke MG, Frusti M, Monaco L, Salgado P, Buso C, Gonzalez CD, Commendatore VF. Glycated Hemoglobin Measurement: Comparison of Three Methods Versus High Performance Liquid Chromatography. J Diabetes Sci Technol. 2022 May;16(3):724-731. doi: 10.1177/1932296821997179. Epub 2021 Mar 9. PMID 33686874
- [Result] van Schaick G, Pot S, Schouten O, den Hartog J, Akeroyd M, van der Hoeven R, Bijleveld W, Abello N, Wuhrer M, Olsthoorn M, Dominguez-Vega E. Evaluating the effect of glycation on lipase activity using boronate affinity chromatography and mass spectrometry. Food Chem. 2023 Sep 30;421:136147. doi: 10.1016/j.foodchem.2023.136147. Epub 2023 Apr 17. PMID 37087987
- [Result] Hoelzel W, Weykamp C, Jeppsson JO, Miedema K, Barr JR, Goodall I, Hoshino T, John WG, Kobold U, Little R, Mosca A, Mauri P, Paroni R, Susanto F, Takei I, Thienpont L, Umemoto M, Wiedmeyer HM; IFCC Working Group on HbA1c Standardization. IFCC reference system for measurement of hemoglobin A1c in human blood and the national standardization schemes in the United States, Japan, and Sweden: a method-comparison study. Clin Chem. 2004 Jan;50(1):166-74. doi: 10.1373/clinchem.2003.024802. PMID 14709644
- [Result] Wu WC, Ma WY, Wei JN, Yu TY, Lin MS, Shih SR, Hua CH, Liao YJ, Chuang LM, Li HY. Serum Glycated Albumin to Guide the Diagnosis of Diabetes Mellitus. PLoS One. 2016 Jan 14;11(1):e0146780. doi: 10.1371/journal.pone.0146780. eCollection 2016. PMID 26765575
- [Result] Atzeni IM, van de Zande SC, Westra J, Zwerver J, Smit AJ, Mulder DJ. The AGE Reader: A non-invasive method to assess long-term tissue damage. Methods. 2022 Jul;203:533-541. doi: 10.1016/j.ymeth.2021.02.016. Epub 2021 Feb 23. PMID 33636313
- [Result] Wolff G, Lin Y, Akbulut C, Brockmeyer M, Parco C, Hoss A, Sokolowski A, Westenfeld R, Kelm M, Roden M, Schlesinger S, Kuss O. Meta-analysed numbers needed to treat of novel antidiabetic drugs for cardiovascular outcomes. ESC Heart Fail. 2023 Feb;10(1):552-567. doi: 10.1002/ehf2.14213. Epub 2022 Nov 7. PMID 36337026